CLINICAL TRIAL: NCT00726557
Title: Quality Assurance of HCV-therapy With PegIntron® Plus Rebetol® in Drug-substituted Patients - SUPPORT Project Post-Marketing Surveillance Study
Brief Title: Post-marketing Surveillance Study of Ex-intravenous Drug Abusers With Chronic Hepatitis C Treated With PegIntron Plus Rebetol (P04408/MK-4031-261)
Acronym: SUPPORT
Status: Completed | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: P04408
Record Dates: First submitted 2008-07-30; First posted 2008-08-01 (Estimated); Results first posted 2010-05-17 (Estimated); Last update posted 2015-10-09 (Estimated); Status verified 2015-10

CONDITIONS: Hepatitis C, Chronic; Substance Abuse, Intravenous
MeSH Terms: conditions — Hepatitis C, Chronic; Substance Abuse, Intravenous | interventions — peginterferon alfa-2b; Ribavirin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PegIntron + Rebetol: There will be a distinction between the patients depending on the type of substitution drug used (secondary parameters).
  Interventions: Biological: PegIntron (pegylated interferon alfa-2b; SCH 54031); Drug: Rebetol (ribavirin; SCH 18908)

INTERVENTIONS:
Biological: PegIntron (pegylated interferon alfa-2b; SCH 54031) — PegIntron 1.5 μg/kg/week administered for a minimum of 12 weeks. Patients who achieve early virologic response at Treatment Week 12, will continue PegIntron therapy for a total of 24 weeks for subjects infected with HCV genotype 2 or 3, and for a total of 48 weeks for subjects infected with HCV genotype 1 or 4
  Other Names: SCH 54031
Drug: Rebetol (ribavirin; SCH 18908) — Rebetol administered at 10.6 mg/kg/day for a minimum of 12 weeks. Patients who achieve early virologic response at Treatment Week 12, will continue Rebetol therapy for a total of 24 weeks for subjects infected with HCV genotype 2 or 3, and for a total of 48 weeks for subjects infected with HCV genotype 1 or 4
  Other Names: SCH 18908

SUMMARY:
Previous intravenous drug abusers with chronic hepatitis C who are under substitution therapy (buprenorphine, methadone) will be treated with PegIntron and Rebetol according to the approved European labeling. The study will assess the tolerability, safety and efficacy of the treatment with PegIntron plus Rebetol in this study population. The objective of the study is to collect data on the prevalence of the hepatitis C infections in drug-substituted patients. The study will also compare the feasibility of HCV (Hepatitis C Virus) treatment in patients receiving Subutex® vs other drug substitution pharmacotherapies.

ELIGIBILITY:
Inclusion Criteria:

* Treatment-naïve participants or relapsers to interferon monotherapy
* Participants with chronic hepatitis C infection
* At least 18 years of age
* Must meet the following laboratory criteria:

  * Platelets >=100,000/mm^3
  * Neutrophil count >=1,500/mm^3
  * TSH (thyroid stimulating hormone) within normal limits
  * Hemoglobin >=12 g/dL (females); >=13 g/dL (males)
* Ex-intravenous drug abusers who are under stable substitution therapy
* Women of childbearing potential must practice adequate contraception and have a routine pregnancy test performed monthly during treatment and for 7 months post-treatment.
* Sexually-active participants must be practicing acceptable methods of contraception during the treatment and for 7 months post-treatment

Exclusion Criteria:

* Any contraindications specified in the SPC (Summary of Product Characteristics) and approved European labeling
* Hypersensitivity to the active substance or to any interferons or to any of the excipients
* Pregnant women
* Women who are breast-feeding
* Existence of or history of severe psychiatric condition, in particular severe depression, suicidal ideation or suicide attempt
* A history of severe pre-existing cardiac disease, including unstable or uncontrolled cardiac disease in the previous 6 months
* Severe debilitating medical conditions, including participants with chronic renal failure or creatinine clearance <50 mL/min
* Coinfection with HIV (Human Immunodeficiency Virus)
* Autoimmune hepatitis or history of autoimmune disease
* Severe hepatic dysfunction or decompensated cirrhosis of the liver
* Pre-existing thyroid disease unless it can be controlled with conventional therapy
* Epilepsy and/or compromised central nervous system function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Previous intravenous drug abusers with chronic hepatitis C receiving substitution therapy (buprenorphine, methadone or other) at approximately 100 sites in Germany.
Sampling Method: Non-Probability Sample
Enrollment: 246 (Actual)
Dates: Start 2005-10; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- PegIntron + Rebetol: PegIntron 1.5 mcg/kg/week + Rebetol 10.6 mg/kg/day administered for a minimum of 12 weeks. Participants who achieved early virological response at Treatment Week 12 continued to receive therapy for a total of 24 or 48 weeks, depending on genotype.
Period: Overall Study
Arm/Group | PegIntron + Rebetol
Started | 246
Completed | 118 (Completed is defined as those who finished the follow-up period.)
Not Completed | 128
Not completed — Screening failure | 4
Not completed — No end of treatment documentation | 37
Not completed — No follow-up documentation available | 55
Not completed — Treatment less than 3 months | 17
Not completed — Inclusion criteria not met | 15

BASELINE CHARACTERISTICS:
Groups:
- PegIntron + Rebetol: Baseline measures only available for the 118 participants who completed.
Arm/Group | PegIntron + Rebetol
Number analyzed (Participants) | 246
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.64 (8.39)
Sex/Gender, Customized [Number; unit: participants]
  Female | 35
  Male | 83
  Unavailable | 128
Region of Enrollment [Number; unit: participants]
  Germany | 246

OUTCOME MEASURES:

1. Primary Outcome: Number of Drug-substituted Participants Who Achieved Sustained Virological Response (SVR) With PegIntron 1.5 μg/kg/Week and Rebetol (10.6 mg/kg/Day) in Substitution Centers Under Routine Conditions
Description: Participants who achieved SVR (sustained virological response) at the end of treatment (24 weeks for genotypes 2,3 and 48 weeks for genotypes 1,4) were analyzed for sustained response at the end of the follow-up period (24 weeks after end of treatment). SVR is defined as having negative HCV-RNA (hepatitis C virus ribonucleic acid).
Time Frame: End of Follow-up (Week 48 or Week 72, depending on genotype)
Population: Participants who achieved SVR at the end of treatment (24 weeks for genotypes 2,3 and 48 weeks for genotypes 1,4)
Measure: Number; unit: Participants
Groups:
- Participants With Negative HCV-RNA at End of Treatment: End of treatment is 24 weeks for genotypes 2,3 and 48 weeks for genotypes 1,4
Arm/Group | Participants With Negative HCV-RNA at End of Treatment
Number analyzed (Participants) | 101
Participants
  Opioid substitution with methadone (n=52) | 49
  Opioid substitution with levo-methadone (n=13) | 10
  Opioid substitution with buprenorphine (n=26) | 23
  Opioid substitution with other medication (n=1) | 0
  No opioid substitution medication (n=9) | 9

2. Primary Outcome: Number of Participants Who Tolerated Treatment With PegIntron 1.5 mcg/kg/Week + Rebetol 10.6 mg/kg/Week
Description: Tolerability of the treatment was measured by number of participants with complete treatment.
Time Frame: Assessed at the end of treatment
Population: All enrolled participants
Measure: Number; unit: participants
Groups:
- Participants Who Tolerated Treatment: Those who completed treatment.
Arm/Group | Participants Who Tolerated Treatment
Number analyzed (Participants) | 246
participants | 118

ADVERSE EVENTS:
Description: Non-serious adverse events (AEs) were not captured as part of the study database. Nevertheless, at the end of each visit, physicians were asked to state if an AE occurred since the last visit. Therefore, it is possible to show only the total number of AEs, which was 104 in the 118 complete participants and 224 in all 246 enrolled participants.
Arm/Group | PegIntron + Rebetol
Serious Adverse Events (participants affected / at risk) | 4/246
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PegIntron + Rebetol (N=246)
Endocarditis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1)
Convulsion (Nervous system disorders) | 1 (1)
Pregnancy of partner (Social circumstances) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Trial results belong to the Sponsor only, all investigators are not allowed to publish trial results without permission of the Sponsor.